CLINICAL TRIAL: NCT04170244
Title: Longitudinal "Real-World" Changes in Skin Microbial Ecology in Atopic Dermatitis (AD) and Psoriasis (PS) Patients
Brief Title: Skin Microbial Ecology in Atopic Dermatitis
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Lisa Beck, Professor, University of Rochester
Other Study IDs: STUDY00003830
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis; Psoriasis; Healthy
Keywords: staphylococcus, microbiome, atopic dermatitis, cutibacterium
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All subjects will have skin swabs and tape strips (done as part of barrier measurements) collected/banked and adult AD subjects will also have serum banked and a small subset of adult (AD and NA) will undergo skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Atopic Dermatitis: Intervention is whatever Rx the URMC dermatologist thinks is best suited to the subject as part of "real-world" disease management in her clinic.
  1. Ages: 1. 13-65 yrs of age (inclusive), all genders, races and ethnicities 2. Additional 66+ yrs of age group, all genders, races and ethnicities
  Interventions: Other: AD subject visit sampling procedures
- Healthy control: No intervention
  Ages:
  1. 13-65 yrs of age (inclusive), all genders, races and ethnicities
  2. Additional 66+ yrs of age group, all genders, races and ethnicities
  Interventions: Other: Healthy control visit sampling procedures
- Psoriasis: Intervention is whatever Rx the URMC dermatologist thinks is best suited to the subject as part of "real-world" disease management in her clinic. Ages:13-65 yrs of age (inclusive), all genders, races and ethnicities.
  Interventions: Other: PS subject visit sampling procedures

INTERVENTIONS:
Other: AD subject visit sampling procedures — Skin swabs for microbial analysis, Tape stripping and transepidermal water loss measurements (TEWL) with tape stripping (all patients) to assess skin barrier function, blood serum (adults & optional for adolescents), and optional biopsy (adults only)
  Groups: Atopic Dermatitis
Other: PS subject visit sampling procedures — Skin swabs for microbial analysis, Tape stripping and transepidermal water loss measurements (TEWL) with tape stripping (all patients) to assess skin barrier function, and blood serum (optional for all PS subjects)
  Groups: Psoriasis
Other: Healthy control visit sampling procedures — Skin swabs for microbial analysis, Tape stripping and transepidermal water loss measurements (TEWL) with tape stripping (all patients) to assess skin barrier function, blood serum (adults & optional for adolescents), and optional biopsy (adults only)
  Groups: Healthy control

SUMMARY:
Everybody's skin has bacteria that normally lives on it. Previous research has shown that people with eczema (or atopic dermatitis [AD]) have much higher concentrations of a certain bacteria (S. aureus), especially when their disease is active but little is known about the role that this bacteria plays in psoriasis (i.e. disease severity, biomarkers and skin barrier function). The overarching purpose of this longitudinal study is to understand how the abundance of skin S. aureus (and several commensal bacteria) change as a consequence of standard of care treatment in the URMC dermatology clinics. Other assays and biospecimens will also be collected to address a number of questions.

DETAILED DESCRIPTION:
Although the two most common inflammatory skin diseases (AD and Psoriasis) are now quite effectively managed with topical and/or systemic therapies, how this disease improvement is reflected in changes of skin microbial pathogens and commensals is still not well understood. We have several aims.

Aim 1 - Determine how the abundance of S. aureus, other microbes of interest including, but not exclusive to, coagulase-negative Staphylococcus species [CONS], and C. acnes on the skin surface varies as a function of time and/or disease activity in AD, plaque stage psoriasis (PS) and healthy, non-atopics (NA). Aim 2 - Validate whether a biomarker (or panel) identifies subjects with greater S. aureus burden (e.g., abundance). Aim 3 - Identify a biomarker (or panel) that predicts clinical improvement observed in our AD or PS subjects. Aim 4 - Quantify S. aureus virulence factors from skin swabs of all three subject populations. Exploratory Aim 5 - Develop a skin microbial repository (optional) where we will focus on the interplay between S. aureus and other microbes from AD and PS patients, and age- and gender-matched healthy NAs. Exploratory Aim 6 - Develop a repository of skin tape strips for biomarker and protease assays. Exploratory Aim 7 - (optional enrollment) - To identify skin epithelial gene signatures from AD skin that are unique and not found in healthy non- AD, NA control skin samples after they are infected ex vivo with HSV-1. A secondary goal of this work will be to evaluate how Real-World treatment(s) affect these observations.

ELIGIBILITY:
Inclusion Criteria:

* ≥13 to 65 years of age (inclusive) for PS, ≥13 for AD and NA, male or female
* Optional Bx sub study - only adults (18-65 yrs; inclusive only)
* Able to understand protocol and give consent
* Able to keep clinic/study appointments and comply with study related procedures
* Must be able to read, speak, and understand English
* Chronic AD, according to the American Academy of Dermatology (AAD) Consensus Criteria (Eichenfield 2014), that has been present for at least 1 year before the enrollment visit
* Chronic PS, according to the AAD Consensus Criteria (Menter et al 2008 (section 1)), that has been present for at least 1 year before the enrollment visit.
* AD subjects: have active lesions on upper extremities, lower extremities, or trunk and a total disease severity of high moderate-to-severe (EASI ≥12)
* PS subjects: have active lesions on upper extremities, lower extremities, or trunk and a total disease severity of high moderate-to-severe (PASI ≥7)

Exclusion Criteria:

* Unwilling and/or unable to complete informed consent process
* <13 or > 65 years of age for PS, >13 for AD and NA
* AD subjects: disease without upper extremity, lower extremity, or trunk lesions
* AD subjects: total disease severity less than moderate (EASI <12), depending on enrollment
* PS subjects: disease without upper extremity, lower extremity, or trunk lesions
* PS subjects: total disease severity less than moderate (PASI <7), depending on enrollment
* Control subjects: diagnosed with an inflammatory skin disease
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the individual's participation in the study (Ex: HIV infection, autoimmune disease, severe heart failure, Hx of malignancy (other than in situ cervical cancer or basosquamous skin cancer), etc.)
* Recent bacterial, fungal, or viral infection requiring systemic therapies (PO, IV or IM) within the last month.
* Subjects with a history of serious life-threatening reaction to tape or adhesives may be enrolled but cannot undergo Tape stripping procedure and will therefore only have a baseline TEWL measurement.
* (For Skin biopsy substudy only) - Subjects with history of keloid formation or allergy to lidocaine.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The healthy population will be defined as individuals with no personal history of or active case of any atopic disorder (e.g. atopic dermatitis, allergic rhinitis, asthma, hay fever). These patients will be individuals seen in URMC Dermatology clinic for a non-infectious condition that does not affect the skin of the extremities. AD subjects must have moderate-to-severe disease defined as an Eczema Area and Severity Index (EASI) of ≥ 12. The psoriasis subjects will have moderate-to-severe disease defined as a Psoriasis Area and Severity Index of ≥ 7. The healthy controls will be recruited to be age- and gendermatched to those with inflammatory skin diseases. Subjects will be recruited from URMC Dermatology clinics at Red Creek and Collegetown.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Abundance of colony forming units (rCFU/cm^2, and CFU/rCFU) of Staphylococcus aureus (S. aureus) | year 1-7
  The abundance of S. aureus, and other microbes of interest including, but not exclusive to, coagulase-negative Staphylococcus species [CONS], and C. acnes present on the skin surface varies as a function of time and/or disease activity in AD and two control groups, namely plaque stage psoriasis (PS) and healthy, non-atopics (NA).
  Standard culture techniques will be utilized to measure rCFU/cm^2, and qPCR for CFU/rCFU.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided